CLINICAL TRIAL: NCT06704022
Title: Assessing Gut Microbiome Changes Before and After an Oral Nutritional Supplement Intake Using the SIMBA Capsule in Diabetic Participants
Status: Not yet recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Nimble Science Ltd. (Industry)
Collaborators: Alberta Obesity Centre (Unknown)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: NIMCSF276
Record Dates: First submitted 2024-11-20; First posted 2024-11-25 (Actual); Last update posted 2025-08-11 (Actual); Status verified 2025-08

CONDITIONS: Type 2 Diabetes
Keywords: oral nutritional supplement; microbiome; small intestine
MeSH Terms: conditions — Diabetes Mellitus, Type 2 | interventions — Dietary Supplements

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Interventional Arm (Experimental): Ingestion of the ONS
  Interventions: Dietary Supplement: Oral nutritional supplement

INTERVENTIONS:
Dietary Supplement: Oral nutritional supplement — Consumption of the oral nutritional supplement

SUMMARY:
This is a single-arm interventional clinical study, the primary objective is to assess the changes in the small intestinal (SI) metagenomic profile of in diabetic participants from baseline to midpoint and endpoint in response to the ONS intervention. The study population is Type 2 Diabetes (T2D) participants (n=30) who will ingest an Oral Nutritional Supplement (ONS) .

DETAILED DESCRIPTION:
This is a single-arm interventional clinical study, the primary objective is to assess the changes in the small intestinal (SI) metagenomic profile of in diabetic participants from baseline to midpoint and endpoint in response to the ONS intervention. The study population is Type 2 Diabetes (T2D) participants (n=30) who will ingest an Oral Nutritional Supplement (ONS) specifically formulated for T2D participants (Glucerna®). While widely used, and despite a strong scientific rationale for their potential influence on the gut microbiota, the impact of nutritional supplements such as Glucerna® has not yet been tested on the gut microbiome. Understanding their impact on the microbiome can lead to new ways for ONS products to better support metabolic health, and long term glucose sugar control. Given the critical role of the small intestine in T2D, the study utilizes the SIMBA capsule to measure novel changes in the small intestine along with traditional measurements from fecal, saliva and blood.

ELIGIBILITY:
Inclusion Criteria:

1. Aged 40-65 years old at the inclusion of the study, both female and male subjects.
2. Has type 2 diabetes as evidenced by their medical history charts and is able to maintain number of medications, type and dose throughout the duration of the study.
3. Has HbA1c ≥ 6.5% and ≤ 9.5% based on a blood sample collected at the Screening Visit, documented within the past month or referred by a medical doctor.
4. Normal to overweight (BMI 20-29.9).
5. Weight is stable (has maintained current body weight within 3 kg) for the two months prior to the Baseline Visit.
6. Is taking a maximum of 3 oral anti-diabetic drugs, one of which must be Metformin. Other class of medications permitted include: Sulfonylurea, SGLT2 inhibitors, and DPP4 inhibitors.
7. Either a male or a non-pregnant, non-lactating female, at least 6 weeks postpartum prior to the Baseline Visit.
8. Willingness to follow the protocol as described, including consumption of study product per the protocol and completing any forms/questionnaires needed throughout the study.
9. The participant is willing to refrain from taking non-study diabetes-specific oral nutritional formulas over the entire course of the study.
10. Willing to maintain their diet and physical activity levels during the study.
11. Able to swallow a 25mm length and 9mm width sized capsule.
12. At least a four-week washout period between the completion of a previous research study that required ingestion of any study food or drug and their start in the current study. Signed Informed Consent; willing and able to comply with study procedures

Exclusion Criteria:

1. Confirmed type 1 diabetes and/or had a history of diabetic ketoacidosis.
2. Use of exogenous insulin or GLP1 agonists for glucose control.
3. Using diabetes-specific oral nutritional supplements(s), (e.g. Glucerna®, Boost etc.) defined as more than one eating occasion per week within the past 4 weeks (those users who can stop using such products for ≥4 weeks before baseline visit need not be excluded).
4. Follows a non-typical eating pattern such as very low carbohydrate diet (e.g., Adkins diet, ketogenic diet, high protein diet).
5. Has eating disorder, severe dementia or delirium, history of significant neurological or psychiatric disorder, alcoholism, substance abuse or other conditions that may interfere with study product consumption or compliance with study protocol procedures in the opinion of the investigators.
6. Galactosemia and lactose intolerance
7. A chronic disease which in the opinion of the investigator, would adversely affect study safety or outcome. Such as, but not limited to

   * A significant cardiovascular event within 6 months prior to study entry or history of congestive heart failure, per physician evaluation.
   * End-stage organ failure (such as end-stage renal disease) or is post-organ transplant.
   * Current or history of renal disease or on dialysis or severe gastroparesis.
   * Current diagnosed hepatic disease such as liver cirrhosis or late-stage liver fibrosis. Participants with prevalent angina will not be excluded.
8. A chronic, contagious, infectious disease, such as active tuberculosis, Hepatitis C, or HIV.
9. Subject has current active malignant disease or was treated within the last 6 months for cancer, except basal or squamous cell skin carcinoma, prior to enrollment.
10. Taking any herbals, dietary supplements, or medications during the past four weeks prior to baseline visit that could profoundly affect (in the opinion of the principal investigator or site physician) blood glucose, body weight, muscle, metabolism, appetite or microbiome (e.g. orlistat, contrave) (naltrexone/bupropion), Qsymia (phentermine/topiramate), Belviq (lorcaserin), incretin mimetics, other drugs indicated for weight loss, cannabis, glucocorticoids, prebiotics and probiotic supplements). Those users who have stopped using such supplements/ medications for ≥4 weeks prior to baseline need not be excluded).
11. Use of any medications in the week prior to the screening study visit, unless part of regular treatment, that could substantially alter gastrointestinal motor function (e.g., opioids, anticholinergics, GLP-1 analogues); laxative use is allowed if it is kept unchanged in the week prior to the SIMBA capsule ingestion timepoints. Proton pump inhibitors (PPIs) are allowed provided a wash-out period of 48 hours is respected before swallowing the SIMBA capsules and PPI treatment is resumed only 4 hours thereafter.

    - If willing prokinetic use can be discontinued for the study duration, with a washout period of 2 weeks
12. Antibiotic use (except for topical use) ≤ 12 weeks prior to screening. Potential participants may be eligible once a 12-week washout is completed.
13. Current infection (requiring medication and antibiotics), inpatient surgery or received systemic corticosteroid treatment [except for inhaled (includes nasal), topical, and ophthalmic steroids] in the last 3 months.
14. Prior gastrointestinal disease, surgery, or radiation treatment which, in the Investigator's opinion, would interfere with consumption or digestion or absorption of study product, lead to intestinal structuring or obstruction with a risk of capsule non-excretion, including, e.g., achalasia, eosinophilic esophagitis, cancer diagnosis or previous esophageal, gastric, small intestinal, or colonic surgery. Appendectomy or cholecystectomy more than 3 months before the screening visit is acceptable.

    - Diagnosed with Crohn's disease, ulcerative colitis or celiac disease.
15. History of known structural gastrointestinal abnormalities such as structures or fistulas leading to mechanical obstruction.
16. Organic motility disorder, including gastroparesis, intestinal pseudo-obstruction, systemic sclerosis, Ogilvie's syndrome.
17. History of oropharyngeal dysphagia, or other swallowing disorder with a risk of capsule aspiration.
18. History of less than three (3) bowel movements per week. 13) Consumption of probiotic or prebiotic capsule supplements within 1 month prior to screening. Potential participants may be eligible once a 1-month washout is completed.
19. Any prior Fecal Microbiota Transplantation.
20. Colon cleanses/bowel prep for 2 weeks.
21. Clotting or bleeding disorders (the use of Plavix® or a similar anticoagulant drug with no reported difficulty during blood draws will be allowed as per physician's opinion).
22. Has blood or blood-related diseases (e.g. hemophilia, thalassemia, sickle cell disease, hereditary spherocytosis, glucose-6-phosphate dehydrogenase deficiency).
23. Received a blood transfusion within the last 3 weeks.
24. Allergic or intolerant to any ingredient found in the study products.
25. Habitually engages in strenuous exercise (e.g., high intensity aerobic exercise, including heavy physical labor), duration of 1 hour or longer, 3 or more times per week. Potential participants may be eligible to participate if their levels exercise are reduced.
26. Participant is actively enrolled in a weight loss program.
27. Are scheduled for an MRI at any time during the study. Potential participants may be eligible to participate once their MRI procedure is completed.
28. Pregnant or breastfeeding.
29. Planning to become pregnant.

Ages: 40 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2025-09 (Estimated); Primary Completion 2026-08 (Estimated); Study Completion 2026-08 (Estimated)

PRIMARY OUTCOMES:
Primary Outcome | Compared at intervention from baseline, midpoint, to endpoint (completion), an average of 6 weeks
  To assess changes in small intestinal metagenomic profile in Type 2 diabetic participants from baseline to midpoint and endpoint in response to the ONS intervention, as measured using the SIMBA capsule.

SECONDARY OUTCOMES:
Secondary 1 | Compared from baseline, midpoint to endpoint (completion), an average of 6 weeks
  Assess the change in metagenomic profile between the blood, saliva, and stool, of Type 2 diabetic participants in response response to the ONS intervention from baseline, to midpoint and endpoint using the SIMBA capsule.
Secondary 2 | Compared from baseline, midpoint to endpoint (completion), an average of 6 weeks
  Assess the change in metabolomic profile in the saliva blood, stool, and SI of Type 2 diabetic participants in response to the ONS intervention from baseline, to midpoint and endpoint using the SIMBA capsule.
Secondary 3 | Compared from baseline, midpoint to endpoint (completion), an average of 6 weeks
  Assess the microbial composition (superimposability of PLS-DA mapping) of the SI from samples collected by the SIMBA capsule
Secondary 4 | Compared from baseline, midpoint to endpoint (completion), an average of 6 weeks
  To assess changes in self-reported satiety in response to the ONS which will be measured at three timepoints: baseline, midpoint, and endpoint.
Secondary 5 | Compared from baseline, midpoint to endpoint (completion), an average of 6 weeks
  Identify potential metagenomic and metabolomic biomarkers that could predict or correlate with the response to the ONS intervention.
Secondary 6 | Compared from baseline, midpoint to endpoint (completion), an average of 6 weeks
  Assess the impact of the ONS intervention on gut function and overall gastrointestinal health, potentially using additional indicators such as gut permeability or inflammatory markers.

CONTACTS AND LOCATIONS:
Locations (1):
- Nimble Science, Calgary, Alberta, Canada

IPD SHARING:
Plan to Share IPD: No